CLINICAL TRIAL: NCT01365650
Title: Open Label, Three-Way Study to Assess the Absorption and Tolerability of Intranasal Ketorolac Tromethamine and to Assess the Effects of a Single Dose of Oxymetazoline Hydrochloride and Multiple Doses of Fluticasone Propionate on the Absorption and Tolerability of Intranasal Ketorolac Tromethamine in Participants With Allergic Rhinitis
Brief Title: Study to Assess the Absorption and Tolerability of Intranasal Ketorolac Tromethamine and to Assess the Effects of Oxymetazoline Hydrochloride and Fluticasone Propionate on the Absorption and Tolerability of Intranasal Ketorolac Tromethamine in Participants With Allergic Rhinitis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ROX 2007-03
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Results first posted 2015-07-23 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Ketorolac Tromethamine; Oxymetazoline; Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Ketorolac Tromethamine (Experimental)
  Interventions: Drug: Ketorolac Tromethamine
- Oxymetazoline Hydrochloride (Experimental)
  Interventions: Drug: Oxymetazoline Hydrochloride
- Fluticasone Propionate (Experimental)
  Interventions: Drug: Fluticasone Propionate

INTERVENTIONS:
Drug: Ketorolac Tromethamine — Single intranasal dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) on Day 1 of Period 1
  Arms: Ketorolac Tromethamine
Drug: Oxymetazoline Hydrochloride — Single intranasal dose of oxymetazoline hydrochloride followed by a single intranasal dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) 30 minutes later on Day 1 of Period 2
  Arms: Oxymetazoline Hydrochloride
Drug: Fluticasone Propionate — Seven days of treatment with intranasal fluticasone propionate (between Periods 2 and 3) followed by a single intranasal dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) on Day 1 of Period 3
  Arms: Fluticasone Propionate

SUMMARY:
This was an open label, three way study in participants with symptomatic allergic rhinitis. The following 3 treatments were administered to each subject during dosing periods 1, 2 and 3, respectively:

* Treatment A: Single intranasal dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) on Day 1 of Period 1.
* Treatment B: Single intranasal dose of oxymetazoline hydrochloride followed by a single intranasal dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) 30 minutes later on Day 1 of Period 2.
* Treatment C: Seven days of treatment with intranasal fluticasone propionate (between Periods 2 and 3) followed by a single intranasal dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) on Day 1 of Period 3.

Subjects remained resident in the Clinical Unit from Day 1 until the morning of Day 2 in each period and there was a washout period of 2 to 7 days between periods. A post study medical was performed within 7 days of Period 3.

The objectives of this study were:

* To assess the pharmacokinetics (PK) of intranasal ketorolac in participants with symptomatic allergic rhinitis.
* To assess the effects of a single dose of intranasal oxymetazoline hydrochloride on the pharmacokinetics and tolerability of intranasal ketorolac in participants with symptomatic allergic rhinitis.
* To assess the effects of chronic administration of fluticasone propionate on the bioavailability and tolerability of intranasal ketorolac in participants with symptomatic allergic rhinitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female volunteers, aged between 18 and 65 years inclusive
* Participant had a history of allergic rhinitis for which treatment had been required at least 3 days out of 7 within the last 3 months. Subjects who were symptomatic of allergic rhinitis but were not currently using therapy because they had found it ineffective may have been included
* Participant was otherwise considered to exhibit general good health, in the opinion of the Investigator
* Participants may have had known medical conditions that were considered "stable" and not expected to interfere with the study outcome or to be adversely affected by their involvement in the study. This was determined by the Investigator at the time of screening by the following:

  * A pre-study physical examination with no clinically significant abnormalities
  * Vital signs within normal ranges or outside the normal range but not deemed clinically significant in the opinion of the Investigator
  * An electrocardiogram (ECG) with no clinically significant abnormalities
  * Full medical history
* Participant had bilateral patent nasal airways at screening as assessed by the Investigator
* Participant had a body mass index (BMI) between 19 and 29 kg/m2
* Female participants of child bearing potential:

  * Must have had a negative urine pregnancy test prior to entry into the study
  * Must not have been breast feeding
* All female participants of child bearing potential and all male participants with female partners of child bearing potential must have consented to use a medically acceptable method of contraception (oral or implanted contraceptive hormones with combined use of barrier contraception, condom or diaphragm with spermicidal agent, intrauterine device, menopausal [defined as last menstrual period >12 months ago] or surgical sterilization) throughout the study period and for a minimum of 4 weeks or 1 full menstrual cycle prior to inclusion
* Participant must have been able to provide written informed consent
* Participant's pre-study clinical laboratory findings were within normal range or if outside of the normal range not deemed clinically significant in the opinion of the Investigator
* Glomerular filtration rate >75 mL/minute as calculated using the Cockroft-Gault calculation for creatinine clearance

Exclusion Criteria:

* Any known allergy or sensitivity to ketorolac tromethamine, oxymetazoline hydrochloride, fluticasone propionate or formulation ingredients
* Any history of co-existing nasal polyps, NSAID sensitivity and asthma
* Daily use of an intranasal decongestant medication
* Allergic reaction to aspirin or other NSAIDs
* Current upper respiratory tract infection or other respiratory tract condition that could have interfered with the absorption of the nasal spray or with the assessment of AEs
* Use of any non-prescribed drug in the 72 hours prior to study drug administration and during the study. Paracetamol use was not allowed within the 24 hours prior to Day 1 of each period. NSAIDs were restricted for at least 3 days or 5 half-lives, whichever was longer, prior to dosing on Day 1 of Period 1, and must not have been used throughout the study. Current prescribed medications were not discontinued prior to entry into the study or during study participation, unless known to interact with ketorolac as per the product information (injectable)
* Any suspicion of rhinitis medicamentosa (chronic daily use of topical decongestants)
* Use of a monoamine oxidase inhibitor in the 14 days prior to study entry
* Positive serum test for human immunodeficiency virus (HIV) or hepatitis B or C at screening
* Positive serum alcohol test at screening or on entry into the study
* Positive urine drug screen for any non-prescribed drugs of abuse (DOA) at screening or on entry into the study
* Clinically significant abnormality on screening laboratory tests
* History of cocaine use
* Concurrent use of ritonavir or other potent CYP3A4 inducers or inhibitors.
* Blood donation within 30 days of beginning study participation
* Active peptic ulcer disease, gastrointestinal bleeding or perforation, or a history of peptic ulcer disease or gastrointestinal bleeding
* Anemia due to unexplained or known gastrointestinal bleeding
* Renal impairment or a risk for renal failure due to volume depletion.
* History of asthma or any other chronic pulmonary disorder, with the exception of childhood asthma and asymptomatic asthma, which were assessed individually by the Principal Investigator
* Current tobacco use or a past history of smoking > or = 5 pack-years within the last 5 years
* A history of any other clinically significant, unstable medical problem, which in the opinion of the Investigator would have interfered with study participation
* Participation in another investigational drug study within 30 days of study entry, or 5 times the half-life of the investigational drug, whichever was longer
* Positive test for Helicobacter pylori (H. pylori) at screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-12; Primary Completion 2008-02 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln Bynum, MD, Study Director — ICON Developmental Solutions
Locations (1):
- Pain and Anaesthesia Research Clinic/Royal Adelaide Hospital, Adelaide, Australia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: December 18, 2007 through February 15, 2008; Medical Clinic
Pre-assignment Details: After subjects had given their informed consent, subjects were required to pass a screening visit within 3 weeks prior to study drug administration.
Groups:
- Symptomatic Allergic Rhinitis: Treatment A: Single intranasal (i.n.) dose of Ketorolac tromethamine (KT) 30 mg (one 15 mg spray into each nostril) on day 1 of Period 1 followed by a 2-7 day washout interval Treatment B: Single i.n. dose of oxymetazoline hydrochloride (OH) followed 30 minutes later by a single i.n. dose of KT 30 mg (one 15 mg spray into each nostril) of Period 2 followed by a 2-7 day washout interval Treatment C: Seven days of treatment with i.n. fluticasone propionate (between Periods 2 and 3) followed by a single i.n. dose of KT 30 mg (one 15 mg spray into each nostril) on day 1 of Period 3
Period: Treatment A
Arm/Group | Symptomatic Allergic Rhinitis
Started | 24
Completed | 24
Not Completed | 0
Period: Treatment B
Arm/Group | Symptomatic Allergic Rhinitis
Started | 24
Completed | 24
Not Completed | 0
Period: Treatment C
Arm/Group | Symptomatic Allergic Rhinitis
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Treatment A: Single intranasal (i.n.) dose of Ketorolac tromethamine (KT) 30 mg (one 15 mg spray into each nostril) on day 1 of Period 1 followed by a 2-7 day washout interval Treatment B: Single i.n. dose of oxymetazoline hydrochloride (OH) followed 30 minutes later by a single i.n. dose of KT 30 mg (one 15 mg spray into each nostril) of Period 2 followed by a 2-7 day washout interval Treatment C: Seven days of treatment with i.n. fluticasone propionate (between Periods 2 and 3) followed by a single i.n. dose of KT 30 mg (one 15 mg spray into each nostril) on day 1 of Period 3
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.6 (16.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 15
Region of Enrollment [Number; unit: participants]
  Australia | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax (the Maximum Observed Plasma Concentration)
Description: PK analysis by standard model was performed by a pharmacokineticist using model-independent analysis methods in WinNonlin Professional. Actual blood sampling times for ketorolac assay were converted to a time from dosing (elapsed time). Elapsed times were listed by subject for each time, together with individual plasma concentrations of ketorolac.
Time Frame: Blood samples for PK analyses were obtained at pre-dose, 0.25, 0.5, 0.75, 1, 1.5, 2, 4, 6, 8, 12, 15 and 24 hours post administration of ketorolac tromethamine
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Single i.n. Dose of 30 mg Ketorolac Tromethamine: Treatment A: Single i.n. dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) on day 1 of Period 1.
- Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a: Treatment B: Single i.n. dose of oxymetazoline hydrochloride followed by a single i.n. dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) 30 minutes later on Day 1 of Period 2.
- Seven Days of Treatment With i.n. Fluticasone Propionate: Treatment C: Seven days of treatment with i.n. fluticasone propionate (between Periods 2 and 3) followed by a single i.n. dose of 30 mg ketorolac tromethamine (one 15 mg spray into each nostril) on day 1 of Period 3.
Arm/Group | Single i.n. Dose of 30 mg Ketorolac Tromethamine | Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a | Seven Days of Treatment With i.n. Fluticasone Propionate
Number analyzed (Participants) | 24 | 24 | 24
ng/mL | 1630.223 (653.599) | 1729.393 (684.055) | 1617.810 (766.328)

2. Primary Outcome: Tmax (the Time to Maximum Concentration)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Single i.n. Dose of 30 mg Ketorolac Tromethamine | Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a | Seven Days of Treatment With i.n. Fluticasone Propionate
Number analyzed (Participants) | 24 | 24 | 24
hours | 1.000 [0.25 to 2.00] | 1.250 [0.75 to 2.05] | 0.875 [0.25 to 4.00]

3. Primary Outcome: AUC 0-t (the Area Under the Plasma Concentration-time Curve (AUC) From Time Zero to the Last Quantifiable Time Point Post-dose)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Single i.n. Dose of 30 mg Ketorolac Tromethamine | Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a | Seven Days of Treatment With i.n. Fluticasone Propionate
Number analyzed (Participants) | 24 | 24 | 24
ng*h/mL | 9001.8 (4011.2) | 9310.3 (3200.2) | 8794.3 (4188.2)

4. Primary Outcome: AUC 0-∞ (the AUC From Time Zero to Infinity, Where Possible)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Single i.n. Dose of 30 mg Ketorolac Tromethamine | Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a | Seven Days of Treatment With i.n. Fluticasone Propionate
Number analyzed (Participants) | 24 | 24 | 24
ng*h/mL | 9906.9 (4347.0) | 9959.1 (3294.8) | 9445.4 (4308.2)

5. Primary Outcome: t1/2z (the Terminal Half-life, Where Possible)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Single i.n. Dose of 30 mg Ketorolac Tromethamine | Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a | Seven Days of Treatment With i.n. Fluticasone Propionate
Number analyzed (Participants) | 24 | 24 | 24
hours | 5.583 (1.929) | 5.172 (1.582) | 5.216 (1.958)

6. Primary Outcome: MRT (the Mean Residence Time)
Description: as for outcome 1
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Single i.n. Dose of 30 mg Ketorolac Tromethamine | Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a | Seven Days of Treatment With i.n. Fluticasone Propionate
Number analyzed (Participants) | 24 | 24 | 24
hours | 7.241 (2.235) | 6.861 (2.037) | 7.088 (2.488)

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Single i.n. Dose of 30 mg Ketorolac Tromethamine | Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a | Seven Days of Treatment With i.n. Fluticasone Propionate
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 17/24 | 22/24 | 17/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single i.n. Dose of 30 mg Ketorolac Tromethamine (N=24) | Single i.n. Dose of Oxymetazoline Hydrochloride Followed by a (N=24) | Seven Days of Treatment With i.n. Fluticasone Propionate (N=24)
Lacrimation increased (Eye disorders) | 3 (3) | 0 (0) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 1 (1) | 5 (5)
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 18 (18) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No